CLINICAL TRIAL: NCT06930625
Title: A Phase 3 Randomized 3-arm Trial (Double-blind Debio 4126, Placebo Control, and Open-label Debio 4126), to Assess the Efficacy and Safety of Debio 4126, a 12-week Octreotide Formulation, in Patients With Acromegaly Previously Treated With Somatostatin Analogs
Brief Title: A Study to Assess the Efficacy and Safety of Debio 4126 in Participants With Acromegaly Previously Treated With Somatostatin Analogs
Acronym: OXTEND™-03
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Debio 4126-301; 2024-516616-24 (Other: EU CT Number); U1111-1310-8427 (Other: WHO Unique Trial Identifier)
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Acromegaly
Keywords: IGF-1; Growth hormone; Pituitary gland; Gigantism
MeSH Terms: conditions — Acromegaly; Pituitary Diseases; Gigantism

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Arms A and B: Period 1 (Double-blind) and Period 2 (Open-label). Arm C: Open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Debio 4126 (Experimental): During Period 1 (double-blind treatment period), participants will receive an intramuscular (IM) injection of Debio 4126 once every 12 weeks over a total of 36 weeks (3 injections in total). Participants whose acromegaly is not well controlled may receive rescue medication.
  Eligible participants (IGF-1 ≤1x ULN on Week 34) will enter Period 2 on Week 36 and receive an open-label Debio 4126 injection once every 12 weeks over a total of 24 to 60 weeks (between 2 and 5 injections in total). Participants with IGF-1 >1x ULN may receive rescue medication until Week 48, and may become eligible for Period 2 if their IGF-1 is ≤1x ULN.
  Interventions: Drug: Debio 4126
- Arm B: Placebo + Debio 4126 (Placebo Comparator): During Period 1 (double-blind treatment period), participants will receive an IM injection of placebo once every 12 weeks over a total of 36 weeks (3 injections in total). Participants whose acromegaly is not well controlled may receive rescue medication.
  Eligible participants (IGF-1 ≤1x ULN on Week 34) will enter Period 2 on Week 36 and receive an open-label Debio 4126 injection once every 12 weeks over a total of 24 to 60 weeks (between 2 and 5 injections in total). Participants with IGF-1 >1x ULN may receive rescue medication until Week 48, and may become eligible for Period 2 if their IGF-1 is ≤1x ULN.
  Interventions: Drug: Debio 4126; Drug: Placebo
- Arm C: Debio 4126 (Open-Label Treatment Period) (Experimental): During the Treatment Period, participants will receive an IM injection of Debio 4126 once every 12 weeks over a total of between 60 and 96 weeks (between 5 and 8 injections in total).
  Interventions: Drug: Debio 4126

INTERVENTIONS:
Drug: Debio 4126 — IM injection, a 12-week extended-release formulation of octreotide
Drug: Placebo — IM injection of mannitol suspension
  Arms: Arm B: Placebo + Debio 4126

SUMMARY:
The primary purpose of this study is to assess the effect of Debio 4126 in the maintenance of the levels of insulin-like growth factor 1 (IGF-1) ≤1x upper limit of normal (ULN) in the double-blind period (Period 1) in comparison to placebo at week 36.

ELIGIBILITY:
Inclusion criteria

1. Patients ≥18 years of age
2. Patients who are receiving octreotide or lanreotide monotherapy for acromegaly for at least 6 months, at a stable dose for the last 12 weeks.
3. IGF-1 at screening ≤1x ULN
4. Acromegaly diagnosis, defined as per protocol
5. Adequate bone marrow, hepatic and renal function
6. To enter Period 2 (Arms A and B): IGF-1 ≤1x ULN at Week 34, or up to Week 48 when treated with rescue medication
7. Other protocol-defined criteria apply

Exclusion criteria

1. Compression of optic chiasm causing visual defects
2. Symptomatic cholelithiasis or bile duct dilatation
3. Planned cholecystectomy during the trial duration
4. Acute or chronic pancreatitis
5. Pituitary radiotherapy
6. Uncontrolled hypothyroidism
7. Uncontrolled diabetes
8. Pituitary surgery within 6 months before screening or planned on trial
9. Treatment with pasireotide within 6 months prior to screening, pegvisomant or dopamine agonists within 3 months prior to screening
10. Recent or ongoing cardiovascular or thromboembolic diseases including heart failure, myocardial infarction, stroke, certain arrythmias, pulmonary embolism
11. Other protocol-defined criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Double-blind Period: Percentage of Participants With IGF-1 ≤1x ULN | 36 Weeks

SECONDARY OUTCOMES:
Arm C: Percentage of Participants With IGF-1 ≤1x ULN | 36 Weeks
Percent Change From Baseline in IGF-1 Values | Up to 108 Weeks
Percentage of Participants With IGF-1 ≤1x ULN | Up to 108 Weeks
Percentage of Participants With Growth Hormone (GH) Level <1 ng/mL | Up to 108 Weeks
Double-blind Period: Percentage of Participants Who Experienced at Least One Treatment-Emergent Adverse Event (TEAE) | Up to 36 Weeks
Percentage of Participants Who Experienced at Least One TEAE | Up to 113 Weeks
Local Tolerability of Debio 4126 as Assessed by Erythema, Swelling, and Induration at the Injection Site Using Investigator Assessment | Up to 108 Weeks
Local Tolerability of Debio 4126 as Assessed by Pain at Injection Site Based on Pain Visual Analog Scale (VAS) Score | Up to 108 Weeks
Double-blind Period: Percentage of Participants Taking Rescue Medication | Up to 36 Weeks
Trough Plasma Concentration (Ctrough) of Debio 4126 | Up to 96 Weeks

CONTACTS AND LOCATIONS:
Locations (69):
- United States (9):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - Harvard Medical School, Boston, Massachusetts
  - Washington University-School of Medicine, St Louis, Missouri
  - Palm Research Center Inc, Las Vegas, Nevada
  - The Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
- Austria (2):
  - Medical University Graz, Graz
  - Medizinische Universitaet Wien - Division of Endocrinology and Metabolism, Vienna
- UZ Gent, Ghent, Belgium
- Brazil (4):
  - CETI - Centro de Estudos em Terapias Inovadoras, Curitiba
  - Nucleo de Pesquisa e Desenvolvimento de Medicamentos (NPDM), Fortaleza
  - Instituto Estadual do Cérebro Paulo Niemeyer (IECPN), Rio de Janeiro
  - Hospital das Clinicas - University of Sao Paulo Medical School, São Paulo
- University Specialized Hospital for Active Treatment of Endocrinology Akad. lv Penchev EAD, Sofia, Bulgaria
- Denmark (2):
  - Rigshospitalet, Blegdamsvej 9, Copenhagen
  - Zealand University Hospital, Køge
- Estonia (2):
  - East Tallinn Central Hospital, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
- France (6):
  - CHU d'Angers, Angers
  - Hospices Civils de Lyon, Bron
  - APHP - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Assistance Publique Hopitaux de Marseille (AP-HM) - Hopital La Conception, Marseille
  - Hopital Haut-Leveque, Pessac
  - CHU Toulouse - Hôpital Larrey, Toulouse
- Germany (3):
  - Charité Universitätsmedizin Berlin, Berlin
  - Klinikum der Universität München Medizinische Klinik und Poliklinik IV - Zi, Munich
  - Universitätsklinikum Würzburg - Poliklinik I - Endokrinologie u. Diabetolog, Würzburg
- Hungary (3):
  - Semmelweis Egyetem, Belgyogyaszati es Onkologiai Klinika, Budapest
  - Eszak-Pesti Centrumkorhaz-Honvedkorhaz Endokrinologia, Budapest
  - University of Szeged Faculty of Medicine, Szeged
- Israel (4):
  - Bnai Zion Medical Center, Haifa
  - Rambam Health Care Campus, Haifa
  - Rabin Medical Center - Beilinson Campus, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (9):
  - Azienda ospedaliero Universitaria di Ferrara, Ferrara
  - Ospedale Policlinico San Martino IRCCS, Genova
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico Milano, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - AOU Federico II Napoli, Napoli
  - Azienda Ospedale Università di Padova, Padua
  - Fondazione Policlinico Universitario A Gemelli, Roma
  - University of Torino, Torino
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Lithuania (2):
  - Lithuanian Health Science University Hospital Kauno klinikos, Kaunas
  - Vaidotas Urbanavicius Sole Proprietor Enterprise, Vilnius
- Poland (4):
  - Centrum Medyczne Intercor Sp. z o.o., Bydgoszcz
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie, Gliwice
  - Department of Endocrinology, Metabolism and Internal Medicine, Poznan University of Medical Sciences, Poznan
  - Uniwersytecki Szpital Kliniczny we Wroclawiu, Wroclaw
- Romania (3):
  - Institutul National de Endocrinologie "C.I. Parhon", Bucharest
  - Delta Health Care, Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj-Napoca, Cluj-Napoca
- University Clinical Center of Serbia, Belgrade, Serbia
- Narodni endokrinologicky a diabetologicky ustav, Ľubochňa, Slovakia
- Spain (7):
  - Hosiptal Universitario de la Ribera, Alzira
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Germans Trias i Pujol, Barcelona
  - Hospital Ramón y Cajal, Madrid
  - Complexo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville
- Sweden (2):
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala
- United Kingdom (2):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Leeds Teaching Hospitals NHS Trust, Leeds

IPD SHARING:
Plan to Share IPD: No